CLINICAL TRIAL: NCT06346899
Title: The Real-World Effectiveness and Safety of Lanadelumab (Takhzyro) and Icatibant (Firazyr®) for Hereditary Angioedema: An Observational Study in China
Brief Title: A Study of Lanadelumab (Takhzyro) and Icatibant (Firazyr®) in Persons With HAE in China
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-743-4012
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group L: Lanadelumab: Participants with HAE who have used only lanadelumab during the study-level retrospective observation period will be observed retrospectively from the start date of the participant-level overall baseline period until the end of participant-level retrospective observation period.
  Interventions: Other: No intervention
- Group I: Icatibant: Participants with HAE who have used only icatibant during the study-level retrospective observation period will be observed retrospectively from the start date of the participant-level overall baseline period until the end of participant-level retrospective observation period.
  Interventions: Other: No intervention
- Group B: Lanadelumab + Icatibant: Participants with HAE who have used both lanadelumab and icatibant during the study-level retrospective observation period will be observed retrospectively from the start date of the participant-level overall baseline period until the end of participant-level retrospective observation period.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a non-interventional study.

SUMMARY:
The Chinese health authority has approved lanadelumab to prevent Hereditary Angioedema (HAE) attacks in persons of 12 years and older. It has also approved icatibant to treat acute HAE attacks in persons 2 years and older.

One of the main aims of this study is to learn about the number of HAE attacks in 1 month in Chinese persons with HAE during their treatment with lanadelumab. The other main aim is to learn how much time is needed to resolve acute HAE attacks when treated with icatibant. Other aims of this study are to learn more about side effects of lanadelumab and icatibant treatment as well as to collect additional information on the treatment with lanadelumab, such as the dose and how often it needs to be given, reasons for stopping the treatment with lanadelumab and how long it was taken until stopping. Participants will be treated by their doctors according to routine medical practice. Only data already available in the medical records of the participants will be reviewed and collected during this study.

ELIGIBILITY:
Inclusion criteria:

* Chinese participants who have received at least one dose of lanadelumab or icatibant from the lanadelumab NMPA approval date (02-Dec-2020) to the date of the day before the 1st site initiation date.
* Informed consent will be obtained from the participant (and/or a legally authorized representative) prior to including that participant as a study participant and accessing that participant's data, except for cases in which the informed consent can be waived by the site.

Exclusion criteria:

• Participation in other interventional studies involving lanadelumab, icatibant, or any other HAE drug or investigational product on or after the date of the participant's lanadelumab or icatibant initiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese participants who have received at least one dose of lanadelumab or icatibant from the lanadelumab national medical products administration (NMPA) approval date (02-Dec-2020) to the date of the day before the 1st site initiation date.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Monthly Rate of HAE Attacks for Each Lanadelumab-treated Participant During the Lanadelumab Exposure Period | From the first dose of study drug up to approximately 3 years 8 months
  The HAE monthly attack rate is defined as the total number of attacks that occurred when the participant was in a lanadelumab exposure period, divided by the total lanadelumab exposure time (in days), multiplied by 28 days.
Median Time to Complete Attack Resolution for Icatibant Treated Participants | From the first dose of study drug up to approximately 3 years 8 months
  Time to complete attack resolution among icatibant-treated participants during the retrospective observation period is defined as the time between icatibant first injection and the earliest time of complete resolution of symptoms for each attack during the retrospective observation period that was treated with icatibant.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) During Lanadelumab and Icatibant Exposure Period | From the first dose of study drug up to approximately 3 years 8 months
  An AE is any untoward medical occurrence in a participant administered a studied drug and which does not necessarily have to have a causal relationship with the studied drug. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, a new disease or worsening in severity or frequency of a concomitant disease, temporally associated with the use of a studied drug, whether or not the event is considered causally related to the use of the product. An SAE is any untoward medical occurrence that at any dose: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event in the opinion of the healthcare provider, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above.
Dosage of Lanadelumab Among Lanadelumab-treated Participant During the Lanadelumab Exposure Period | From the first dose of study drug up to approximately 3 years 8 months
  Dosage of lanadelumab used during the lanadelumab exposure period will be assessed.
Frequency Administration of Lanadelumab Among Lanadelumab-treated Participant During the Lanadelumab Exposure Period | From the first dose of study drug up to approximately 3 years 8 months
  Frequency administration of lanadelumab among lanadelumab-treated participant during the lanadelumab exposure period will be assessed.
Number of Participants with Reasons of Discontinuation of Lanadelumab During the Lanadelumab Exposure Period | From the first dose of study drug up to approximately 3 years 8 months
  Number of participants with reasons of discontinuation of lanadelumab during the lanadelumab exposure period will be assessed.
Time to Lanadelumab Discontinuation Among Lanadelumab-treated Participant During the Lanadelumab Exposure Period | From the first dose of study drug up to approximately 3 years 8 months
  The time to lanadelumab discontinuation is defined as the time from lanadelumab initiation to the first lanadelumab discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (13):
- China (13):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujan
  - The First Affiliated Hospital ,Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital,Tongji Medical College,Huazhong University of Science & Technology, Wuhan, Hubei
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qianfo Mountain Hospital, Shandong Province, Jinan, Shandong
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Bethune hospital, Taiyuan, Shanxi
  - The Second Affiliated hospital of Xian Jiaotong University, Xian, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - First Affiliated hospital of Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/7a511c1ac845420c??page=1&idFilter=TAK-743-4012